CLINICAL TRIAL: NCT00567320
Title: Efficacy of Varenicline in Methadone-Stabilized Cocaine Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 0702002337; R01DA021264 (NIH); DPMC (Other: NIDA); MIRECC 000000000 (Registry Identifier: Department of Veterans Affairs)
Record Dates: First submitted 2007-12-03; First posted 2007-12-04 (Estimated); Results first posted 2012-04-09 (Estimated); Last update posted 2020-04-02 (Actual); Status verified 2013-01

CONDITIONS: Cocaine Dependence; Nicotine Dependence
Keywords: varenicline
MeSH Terms: conditions — Cocaine-Related Disorders; Tobacco Use Disorder | interventions — Varenicline; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Active Comparator)
  Interventions: Drug: Varenicline
- Sugar Pill or Placebo (Active Comparator): Placebo is compared to active drug varenicline
  Interventions: Drug: Sugar pill or Placebo

INTERVENTIONS:
Drug: Varenicline — Varenicline up to 2 mg a day
  Other Names: Chantix
  Arms: Varenicline
Drug: Sugar pill or Placebo — Placebo
  Other Names: Sugar pill
  Arms: Sugar Pill or Placebo

SUMMARY:
Cocaine addiction continues to be an important public health problem in the US with a significant cost to the individual and society. Among substance abusers, cocaine use has been recognized as a significant problem especially in methadone-maintenance patients. In several studies, rates of cocaine use have been reported to range from 30 to over 60 percent of those in methadone maintenance programs (Condelli et al. 1991; Hunt et al. 1984; Kidorf and Stitzer 1993; Kosten et al. 1988). In these patients, cocaine use seems to be a predictor of poor clinical outcome (Hartel et al. 1995; Kosten et al. 1987a). The development of effective pharmacotherapies for cocaine use disorders, especially in the opioid-dependent population is of great importance. Unfortunately, such effective pharmacotherapies do not exist.

1. To determine the safety and tolerability of varenicline in cocaine-using methadone-stabilized subjects.
2. To determine if varenicline is efficacious in reducing cocaine-use in methadone-stabilized subjects.

DETAILED DESCRIPTION:
For this pilot study, we hope to recruit a total of 40 subjects, with 20 subjects in the varenicline group, and 20 into the placebo-control group. Assuming significant findings, these data will enable us to estimate a possible effect size for carrying-out a larger study. For preliminary analysis as a prelude to planning larger controlled studies, we will clinically require an effect size of 20% differences in the rates of cocaine positive urines or of self-reported cocaine use between the active medication and placebo groups. We will not adjust for these multiple comparisons to the placebo group since this is a pilot study, and use two-tailed significance level of 0.05 when we employ repeated measures analysis of variance (ANOVA) or Hierarchical Linear Modeling (HLM,see below) for statistical analysis over the 16-week study period.

An Amendment was made and a new Updated consent form to include new FDA findings for study medication Varenicline." Varenicline may also cause changes in behavior, agitation, depressed mood, suicidal ideation and suicidal behavior." Currently we have 30 subjects who have completed this study. This study is suspended due to these new concerns, Department of Veterans Affairs and the P.I. James Poling agreed.

Study has been published. (April 2011)

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 18 and 55 years old will be eligible for this study. Females must not be pregnant as determined by pregnancy screening, nor breast feeding, and must be using acceptable birth control methods during study participation.
* Current opioid dependence as evidenced by documentation of prior treatment for opioid dependence or signs of withdrawal, self-reported history of opioid dependence for consecutive 12 month period and a positive urine for opiates.
* Subjects must fulfill Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for opioid dependence.
* Subjects must have a history of cocaine use, with a reported street cocaine use of a minimum of 1/2 gram during the preceding 30 days.
* Subjects must meet DSM-IV criteria for cocaine dependence or abuse, and have laboratory confirmation of recent cocaine use (positive urine for cocaine) during the month prior to study entry.
* Subjects must be treatment-seekers for opioid and cocaine use.
* Subjects must have smoked at least 10 cigarette per day for at least one year. Varenicline's safety has only been studied in smokers.

Exclusion Criteria:

* History of heart disease, left ventricular hypertrophy, ischemic ECG changes, chest pain, arrhythmia, hypertension.
* History of severe renal or hepatic diseases.
* History of psychosis, schizophrenia, bipolar or major depressive disorder.
* History of seizure disorder.
* Current diagnosis of alcohol, benzodiazepine and other drug abuse or dependence (other than opiates, cocaine, and nicotine).
* Current use of over-the-counter or prescription psychoactive drugs (antidepressant, anxiolytics, antipsychotics, mood stabilizers, psychostimulants).
* Liver function tests (ALT or AST) greater than 3 times normal.
* Known allergy to varenicline or methadone.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2007-03; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Poling, Ph.D., Principal Investigator — Yale University
Locations (1):
- Veterans Hopsital, West Haven, Connecticut, United States

REFERENCES:
- [Result] Poling J, Rounsaville B, Gonsai K, Severino K, Sofuoglu M. The safety and efficacy of varenicline in cocaine using smokers maintained on methadone: a pilot study. Am J Addict. 2010 Sep-Oct;19(5):401-8. doi: 10.1111/j.1521-0391.2010.00066.x. PMID 20716302
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273

RESULTS

PARTICIPANT FLOW:
Groups:
- Varenicline: Varenicline 2 mg per day.
- Placebo: This is the Placebo condition
Period: Overall Study
Arm/Group | Varenicline | Placebo
Started | 13 | 18
Completed | 13 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 13 | 18 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (12) | 34.4 (12) | 35.45 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 11 | 14 | 25
Region of Enrollment [Number; unit: participants]
  United States | 13 | 18 | 31

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Cocaine Positive Urine Tests Per Week
Description: Urine samples were obtained thrice-weekly and analyzed for the presence of cocaine metabolites. Levels that exceeded 300 ng / ml on each individual urine test were considered positive. The primary outcome measure was the proportions of positive cocaine urine results per week that was calculated by using the total number of completed tests as the denominator and the total number of positive tests for that week as the numerator. This data was subjected to Hierarchical Linear Modeling (HLM) analysis using a total of 13 longitudinal results that included a baseline result (Week 0).
Time Frame: Weekly Measures over 12 weeks
Population: Intention to treat analysis of all subjects receiving medication
Measure: Mean (Standard Deviation); unit: Proportion of cocaine positive
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 13 | 16
Proportion of cocaine positive | .57 (.05) | .58 (.05)
Statistical Analysis 1: Comparison: Varenicline vs Placebo; HLM analysis of % of Cocaine Positive Urines per week over 12 weeks. Subjects were used as a Random variable, with medication dosing set to 'Fixed'; Test type: Superiority or Other; p = 0.84, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/16
Other Adverse Events (participants affected / at risk) | 0/13 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No